CLINICAL TRIAL: NCT04493593
Title: Internet-delivered CBT Intervention (Space for Sleep) for Insomnia: Pilot and Feasibility Study in a Routine Care Setting
Brief Title: Internet-delivered CBT-I (Space for Sleep): Pilot and Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silver Cloud Health (Other)
Collaborators: Berkshire Healthcare NHS Foundation Trust (Other); University of Dublin, Trinity College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sleep_IAPT
Record Dates: First submitted 2020-07-09; First posted 2020-07-30 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Insomnia
Keywords: insomnia; online interventions; CBT; IAPT; depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Space for Sleep Group (Experimental): SilverCloud internet-delivered CBT intervention for Insomnia
  Interventions: Behavioral: SilverCloud

INTERVENTIONS:
Behavioral: SilverCloud — 'Space for Sleep' is a seven-module online CBT-based intervention for sleep. The structure and content of the programme modules follow evidence-based CBT principles for insomnia. Each module is structured to incorporate introductory quizzes. videos, informational content, interactive activities, as well as homework suggestions and summaries. In addition, personal stories and accounts from other users are incorporated into the presentation of the material.
  As per normal service provision, each participant will be assigned a clinician (PWP) who will monitor participants' progress through the program. Every one to two weeks, the PWP will login and review participants' progress, leaving feedback for them and responding to the work they have completed.

SUMMARY:
The principal objective of the study is to assess the feasibility and preliminary efficacy of an online-delivered CBT-I intervention for those with insomnia or reporting sleep difficulties. The program will be offered to service users of IAPT to establish criteria for the planning of a future large scale RCT study.

DETAILED DESCRIPTION:
Meta-analytic evidence have shown that internet-delivered CBT-I works at improving insomnia severity, sleep efficiency, subjective sleep quality, wake after sleep onset, sleep onset latency, total sleep time, and number of nocturnal awakenings at post-treatment (Zachariae et al., 2016). Furthermore, these interventions have also been shown efficacious in decreasing depressive symptoms (Christensen et al., 2016).

However, no studies have explored the effects of internet-delivered CBT-I in routine care settings and all of them recruited a self-selected sample, which limits the generalizability of the results. In this sense, the present study is a first step to assess the feasibility and preliminary efficacy of internet-delivered CBT-I in a real-world setting: the Improving Access to Psychological Therapies (IAPT) program, National Health service, England.

The IAPT program is part of a stepped care model that principally addresses depression and anxiety in the population (Clark, 2011). It sees over a million users per year and delivers both low-intensity (e.g. internet-delivered CBT for depression and anxiety disorders; group wellbeing courses, bibliography) and high-intensity (e.g. counseling for depression, face-to-face CBT for depression and anxiety) services (Clark, 2011).

Within IAPT, SilverCloud Health as a global leader in the development and implementation of internet-delivered interventions for mental health, wellbeing and long-term condition management, has supported patients at a low-intensity level (i.e. Step 2) over the past 5 years. SilverCloud has recently developed an intervention for insomnia that will form part of the overall mental health care suite of programs that include interventions for depression and anxiety disorders. The outcomes of these online interventions have been equal to other low-intensity interventions used within IAPT. The current study seeks to pilot the newly developed CBT-I intervention to assess its initial clinical impact and to establish criteria for the planning of a future large scale RCT study.

Objective As part of service evaluation, patients at Berkshire NHS Foundation trust availed of the Space for Sleep program. The current study seeks to carry out research on the progress of these patients, assessing the program's initial clinical impact and to establish criteria for the planning of a future large scale RCT study.

Specific research questions will be the following:

* Can Space for Sleep achieve positive clinical outcomes for patients?
* What are the levels of satisfaction and acceptance of users with the intervention?
* What are the levels of usage of the intervention?

Design Moving from service evaluation to an open feasibility trial design to examine the potential clinical impact of an online CBT intervention for insomnia disorder (ID).

Hypotheses SilverCloud online interventions for mental health have proved highly successful. The investigators anticipate that the current intervention for ID will show preliminary effectiveness at post-treatment in terms of greater sleep efficiency and significant reductions in symptoms of insomnia and co-morbid depression and anxiety.

Study Setting The study will be conducted within Berkshire Healthcare NHS Foundation Trust through Talking Therapies, an NHS IAPT provider that serves a population of 900,000 across 7 Clinical Commissioning Groups (CCGs), all of which are demographically and economically diverse, ranging from rural West Berkshire to urban commuter towns close to London. Talking Therapies aims to provide an easily accessible and clinically effective service for those within the community who suffer from sleep disorders. Those wishing to access the service can do so through self-referral, GP referral or referral from allied services. If suitable, clients are offered treatment either at Step 2 or Step 3 based on their need. Step 2 services include low-intensity CBT-based treatments such as self-help, iCBT and group treatment, supported by trained psychological wellbeing practitioners (PWP).

Recruitment procedures The aim is to recruit 35 patients as part of service evaluation. A 50% uplift is added to buffer against the effects of dropout/missing data. Therefore, a total of 52 participants will be included in the study. Patients who are already using the program as part of the service evaluation will be provided with an information sheet and asked if they wish to retrospective consent to for their data to be part of the research trial.

For those who will be recruited into the research, firstly, individuals are given an initial assessment by phone with a PWP clinician at Berkshire IAPT service as per normal service provision. The assessment determines if an individual meets the eligibility criteria and a diagnosis of sleep disorder will be advised by the PWP. The PWP then describes the trial and invites the client to participate. Those interested will receive an email with information detailing the study and a link to the consent form to give consent by means of a digital signature. Upon giving consent, participants complete the primary and secondary outcomes for the study online. PWPs will reiterate details of the research and the program, describing what is involved and the importance of their participation in the trial. Participants receive an email informing them on how to proceed.

All participants are informed that they are free to withdraw if they no longer wish to take part in the trial. In this case, they will be removed from the trial and they will be offered treatment as usual.

Support during treatment Each participant will be assigned a PWP clinician who will monitor participants' progress throughout the trial. Once assigned to the active treatment condition the participant will receive a message from their PWP clinician at their first login. This message welcomes them to the program, highlights aspects of the program, and encourages them in use of the program. Over the course of the 8-week supported intervention, on 6 separate occasions the PWP will login and review participants progress, leaving feedback for them and responding to the work they have completed. The basic share level allows supporters to view users' goals for the week; key messages and progress points. If users wish to share more with their supporter, they can share journal entries. Each supporter will provide post-session feedback of between 10 and 15 minutes per participant per session, over the eight-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Reporting difficulty getting to sleep and/or staying asleep as their primary presentation
* Suitability for an internet intervention (i.e. willingness to engage on the iCBT intervention, ability to read English, access internet, the capacity and willingness to consent)
* No suicidal or self-harm risk and no specific communication needs.

Exclusion Criteria:

* Score above 0 on PHQ-9 question 9
* Diagnosed psychotic illness
* Currently on psychological or pharmacological treatment for sleep disorder
* Alcohol or drug misuse
* Previous diagnosis of an organic mental health disorder,
* Have an unstable medication regimen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Changes in insomnia severity (as measured by the Insomnia Severity Index, ISI) | Baseline - Immediately after the intervention
  The 7-item ISI (Yang, Morin, Schaefer, & Wallenstein, 2009) provides a quantitative index of overall sleep impairment. Participants rate the severity of sleep problems (e.g. problems with sleep onset, sleep maintenance, and early morning awakening), interference with daytime functioning, how noticeable the impairment is to others, distress or concern caused by the sleep problem(s), as well as satisfaction with the current sleep pattern on a 5-point Likert scale. Scores range from 0-28, with higher scores indicating more severe insomnia. The ISI has been shown to be a valid and reliable measure that is sensitive to changes in treatment studies (Bastien, Vallières, & Morin, 2001; Thorndike et al., 2011).
Changes in average sleep efficiency (i.e. total time spent asleep divided by the total time spent in bed in a given day) | Baseline - Immediately after the intervention
  Sleep efficiency is the result of total time spent asleep divided by the total time spent in bed and multiplied by 100. Participants will be encouraged to complete a sleep diary which is available to them as a tool on the platform. They will be encouraged to complete this throughout treatment and will be prompted to do so upon their daily login. Data from the first and last week will be used as pre- and post-treatment measurements. Sleep efficiency of 85% or above is considered normal, with really good efficiency being 90% or above.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline - Immediately after the intervention
  The PHQ-9 (Kroenke, Spitzer, & Williams, 2001; Spitzer, Kroenke, & Williams, 1999) is a self-report measure of depression that has been widely used in research and is a regular screening measure utilised in primary care and hospital settings. The PHQ-9 items reflect the diagnostic criteria for depression outlined by the DSM-V (American Psychiatric Association, 2013). Summary scores range from 0 to 27, where larger scores reflect a greater severity of depressive symptoms. The PHQ 9 has been found to discriminate well between depressed and non-depressed individuals using the cut-off total score ≥ 10, with good sensitivity (88.0%), specificity (88.0%) and reliability (Kroenke et al., 2001; Spitzer et al., 1999).
Generalized Anxiety Disorder-7 (GAD-7) | Baseline - Immediately after the intervention
  The GAD-7 (Spitzer, Kroenke, Williams, & Löwe, 2006) comprises 7 items measuring symptoms and severity of anxiety based on the DSM-V (American Psychiatric Association, 2013) diagnostic criteria for GAD. The measure has good internal consistency (α = .92) and good convergent validity with other anxiety scales (Spitzer et al., 2006). Higher scores indicate greater severity of symptoms. The GAD-7 has increasingly been used in large-scale studies as a generic measure of change in anxiety symptomatology, using a cut-off score of 8 (Richards & Suckling, 2009).
Work and Social Adjustment Scale (WSAS) | Baseline - Immediately after the intervention
  The WSAS (Mundt, Marks, Shear, & Greist, 2002) is a simple and reliable (α >.75) 5-item self-report measure of impaired functioning, which provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships. Scores range from 0 to 40, with higher score indicating poorer adjustment. WSAS has demonstrated good internal reliability (α = 0.82) (Zahra et al., 2014).
Patient Experience Questionnaire (PEQ) | Immediately after the intervention
  This will be used to assess patient experience and satisfaction. This questionnaire forms a part of the IAPT minimum data set and is a national requirement in the UK. The PEQ contains several quantitative questions and open-ended questions that are used to assess participant's views and satisfaction with service provision.
Acceptability of the modules | Immediately after each module of the intervention
  Each module contains 5 questions that assess the perceived usefulness and acceptability of the module. 4 questions are rated in a 4-point Likert scale ranging from 1 (strongly agreee) to 4 (strongly disagree) where the users report their level of agreement, while the last question is an open box where the users may include additional feedback about the module. Lower scores are indicative of higher acceptability of the module.
Time spent in the platform | During the intervention
  This metric corresponds to the combination of the time spent in each session (in minutes) from the first to the last log-in.
Number of sessions | During the intervention
  This metrics relates to the number of times (log-ins) the user accessed the program.
Number of Activities | During the intervention
  This metric is calculated by counting all the times users interacted actively with the platform, that is, every time that they completed a journal entry, used an interactive tool, or downloaded or played relaxation audios.
Percentage of the Program Viewed | During the intervention
  This metric refers to the percentage of the total program content that the user has gone through.
Number of Reviews | During the intervention
  This metric refers to the number of messages that the supporter sent to the user to encourage use of the platform while providing feedback about the progress from the last review.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, Study Director — SilverCloud Health; Sarah Sollesse, Principal Investigator — Berkshire NHS Foundation Trust
Locations (1):
- Berkshire NHS Foundation Trust, Bracknell, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Christensen H, Batterham PJ, Gosling JA, Ritterband LM, Griffiths KM, Thorndike FP, Glozier N, O'Dea B, Hickie IB, Mackinnon AJ. Effectiveness of an online insomnia program (SHUTi) for prevention of depressive episodes (the GoodNight Study): a randomised controlled trial. Lancet Psychiatry. 2016 Apr;3(4):333-41. doi: 10.1016/S2215-0366(15)00536-2. Epub 2016 Jan 28. PMID 26827250
- [Background] Clark DM. Implementing NICE guidelines for the psychological treatment of depression and anxiety disorders: the IAPT experience. Int Rev Psychiatry. 2011 Aug;23(4):318-27. doi: 10.3109/09540261.2011.606803. PMID 22026487
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Richards DA, Suckling R. Improving access to psychological therapies: phase IV prospective cohort study. Br J Clin Psychol. 2009 Nov;48(Pt 4):377-96. doi: 10.1348/014466509X405178. Epub 2009 Feb 9. PMID 19208291
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Thorndike FP, Ritterband LM, Saylor DK, Magee JC, Gonder-Frederick LA, Morin CM. Validation of the insomnia severity index as a web-based measure. Behav Sleep Med. 2011;9(4):216-23. doi: 10.1080/15402002.2011.606766. PMID 22003975
- [Background] Yang M, Morin CM, Schaefer K, Wallenstein GV. Interpreting score differences in the Insomnia Severity Index: using health-related outcomes to define the minimally important difference. Curr Med Res Opin. 2009 Oct;25(10):2487-94. doi: 10.1185/03007990903167415. PMID 19689221
- [Background] Zachariae R, Lyby MS, Ritterband LM, O'Toole MS. Efficacy of internet-delivered cognitive-behavioral therapy for insomnia - A systematic review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2016 Dec;30:1-10. doi: 10.1016/j.smrv.2015.10.004. Epub 2015 Oct 24. PMID 26615572
- [Background] Zahra D, Qureshi A, Henley W, Taylor R, Quinn C, Pooler J, Hardy G, Newbold A, Byng R. The work and social adjustment scale: reliability, sensitivity and value. Int J Psychiatry Clin Pract. 2014 Jun;18(2):131-8. doi: 10.3109/13651501.2014.894072. Epub 2014 Mar 16. PMID 24527886